CLINICAL TRIAL: NCT05938647
Title: Characteristics of Patients With Severe Dengue Admitted in Critical Care Units at Villavicencio, Colombia. A Retrospective Observational Trial.
Brief Title: Severe Dengue in Critical Care at Villavicencio, Colombia.
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Principal investigator, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2023_02_DENGUE
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Severe Dengue
MeSH Terms: conditions — Severe Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dengue hemorrhagic fever group 3: Risk factor (severity 3): no diagnostic or therapeutic intervention; the characteristics of participants will be analyzed by demographics, severity, laboratory results, fluids accumulation, and outcomes.
  Interventions: Other: Risk factor: group 3
- DHF group 4 (DSS);: Risk factor (group 4): no diagnostic or therapeutic intervention; the characteristics of participants will be analyzed by demographics, severity, laboratory results, fluids accumulation, and outcomes.
  Interventions: Other: Risk factor: group 4

INTERVENTIONS:
Other: Risk factor: group 3 — Severe dengue, no shock. No diagnostic or therapeutic intervention; the characteristics of participants will be analyzed by demographics, severity, laboratory results, fluids accumulation, and outcomes.
  Groups: Dengue hemorrhagic fever group 3
Other: Risk factor: group 4 — Dengue shock syndrome. No diagnostic or therapeutic intervention; the characteristics of participants will be analyzed by demographics, severity, laboratory results, fluids accumulation, and outcomes
  Groups: DHF group 4 (DSS);

SUMMARY:
Severe dengue is a cause of admission to critical care, especially in pediatric cases, and during epidemic outbreaks. Fluid support is basically the therapy offered, due to a scarcity of antiviral or immunological options to modulate the disease. Dengue is an endemic condition in tropical and subtropical regions as Villavicencio, and local ICUs provide care to the adult and pediatric population from the city and distant surrounding areas. National and international agencies' clinical guidelines have standard recommendations for the therapy of dengue shock syndrome (DSS), but data about performance is not available. Severity, organ dysfunction, hemorrhagic events, and capillary leak are predictors for decease. There are several epidemiological trials about dengue in the region, although publications about the characteristics of patients in ICU are nearly null. Currently, there is enough human resources and technology in ICU to provide an optimal care in cases of severe dengue. There is a need to recognize most appropriate strategies for the treatment of the disease, and their results, to adjust and provide better outcomes.

The aim of the study is to analyze the characteristics of patients with severe dengue admitted to the intensive care unit, to contribute to knowledge and better understanding of the disease in a specific clinical environment.

An observational retrospective study will be designed by the analysis of the ICU database of hospitals from Villavicencio, Colombia, since January to May 2023. The records of patients admitted with a diagnose of severe dengue will be exported to Excel for reviewing and debugging. Demographic information, laboratory results, severity scores, and outcomes will be examined. Categorical variables will be described by frequency and proportion; quantitative variables will be defined in a central and dispersion distribution. Chi-square and Mann-Whitney U test will be used to compare, according to the characteristics of the outcome.

It will be a pioneer study at this region, and it is necessary to determine the characteristics of patients admitted to the intensive care unit, the care provided, and the results of the treatment.

DETAILED DESCRIPTION:
Dengue is an endemic viral infection in tropical and subtropical regions like Colombia, with epidemic outbreaks every three years, with severity especially in pediatric cases. Clinical symptoms, and signs are the fundamental strategies for the diagnosis, although they are not explicit for the disease, so it can be undetected. No specific antiviral therapy is available yet.

An increase in the vascular permeability is observed in severe cases. Some viral, and individual characteristics are recognized as risk factors for severity. Viral serotype, secondary infection, comorbidities, and individual genetic host factors predispose to a hyperinflammatory stage and increased response to the infection.

About 5% of severe cases have risk of mortality. Early detection of warning signs, hydration and appropriate care is crucial to prevent decease, and severe cases require proper attention in an ICU for monitoring, fluid restoration, and support of organ dysfunction.

Aggressive fluid therapy is proposed by national and international health organisms, based and limited trials. Crystalloids initial boluses and high fluid therapy are recommended to counter capillary leakage. It involves a risk of fluid overload with chances of secondary injury as pulmonary edema, tissue hypoperfusion, and organ disfunction.

Personalized monitoring of fluid therapy is necessary to achieve the goals of therapy, replacing fluid loss, but reducing timely the accumulated balance. ICU admission offers the opportunity to accomplish such a goal by adjusting the clinical practice guidelines to individual and dynamic needs, based in scientific evidence.

Several publications have evaluated strategies of fluid therapy in sepsis and shock, considering four overlapping phases (ROSE): resuscitation; optimization; stabilization; and evacuation. None of the studies have evaluated patients with dengue.

Determining the characteristics of patients admitted to the ICU by severe dengue, will provide essential information of severity, the therapy provided, the type of support delivered, and the outcomes attained. It will improve the knowledge about the accomplishment of clinical practice guidelines and its results.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at a critical care unit with a diagnose of dengue either clinical or by a positive serology or molecular diagnostic methods.

Exclusion Criteria:

* Patients with a post admission diagnosis different than dengue either clinical or by a negative serology.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants in the trial are those patients treated in a critical care unit for dengue during the period of study, according to the registers of admission in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Number of deaths | 30-days
  Hospital death

SECONDARY OUTCOMES:
Amount of fluid accumulation | 5 days
  Daily positive fluid balance

OTHER OUTCOMES:
Number of ICU days | 30 days
  Length of ICU stay
Number of hospital days | 30-days
  Length of hospitalization
Number of participants with mechanical ventilation | 30-days
  Need of mechanical ventilation
Number of days in mechanical ventilation | 30-days
  Length of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez-Gutierrez, MD, Principal Investigator — Cooperative University of Colombia
Locations (2):
- Colombia (2):
  - Clinica Primavera, Villavicencio, Meta Department
  - Hospital Departamental de Villavicencio, Villavicencio, Meta Department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen CM, Chan KS, Yu WL, Cheng KC, Chao HC, Yeh CY, Lai CC. The outcomes of patients with severe dengue admitted to intensive care units. Medicine (Baltimore). 2016 Aug;95(31):e4376. doi: 10.1097/MD.0000000000004376. PMID 27495047
- [Result] Gupta S, Gupta M, Kashyap JR, Arora SK. Early cardiovascular involvement in dengue fever: A prospective study with two-dimensional speckle tracking echocardiography. Trop Doct. 2022 Apr;52(2):285-292. doi: 10.1177/00494755221076686. Epub 2022 Jan 31. PMID 35098804
- [Result] Madanayake P, Jayawardena A, Wijekoon SL, Perera N, Wanigasuriya J. Fluid requirement in adult dengue haemorrhagic fever patients during the critical phase of the illness: an observational study. BMC Infect Dis. 2021 Mar 20;21(1):286. doi: 10.1186/s12879-021-05971-6. PMID 33743614
- [Result] McBride A, Vuong NL, Van Hao N, Huy NQ, Chanh HQ, Chau NTX, Nguyet NM, Ming DK, Ngoc NT, Nhat PTH, Phong NT, Tai LTH, Tho PV, Trung DT, Tam DTH, Trieu HT, Geskus RB, Llewelyn MJ, Thwaites CL, Yacoub S. A modified Sequential Organ Failure Assessment score for dengue: development, evaluation and proposal for use in clinical trials. BMC Infect Dis. 2022 Sep 3;22(1):722. doi: 10.1186/s12879-022-07705-8. PMID 36057771
- [Result] Rosenberger KD, Alexander N, Martinez E, Lum LCS, Dempfle CE, Junghanss T, Wills B, Jaenisch T; DENCO Clinical Study Group. Severe dengue categories as research endpoints-Results from a prospective observational study in hospitalised dengue patients. PLoS Negl Trop Dis. 2020 Mar 4;14(3):e0008076. doi: 10.1371/journal.pntd.0008076. eCollection 2020 Mar. PMID 32130212
- [Result] Sachdev A, Pathak D, Gupta N, Simalti A, Gupta D, Gupta S, Chugh P. Early Predictors of Mortality in Children with Severe Dengue Fever: A Prospective Study. Pediatr Infect Dis J. 2021 Sep 1;40(9):797-801. doi: 10.1097/INF.0000000000003179. PMID 34321449
- [Result] Sengupta SP, Nugurwar A, Jaju R, Khandheria BK. Left ventricular myocardial performance in patients with dengue hemorrhagic fever and thrombocytopenia as assessed by two-dimensional speckle tracking echocardiography. Indian Heart J. 2013 May-Jun;65(3):276-82. doi: 10.1016/j.ihj.2013.04.017. Epub 2013 Apr 9. PMID 23809381
- [Result] Suwarto S, Nainggolan L, Sinto R, Effendi B, Ibrahim E, Suryamin M, Sasmono RT. Dengue score: a proposed diagnostic predictor for pleural effusion and/or ascites in adults with dengue infection. BMC Infect Dis. 2016 Jul 8;16:322. doi: 10.1186/s12879-016-1671-3. PMID 27391122
- [Result] Swamy AM, Mahesh PY, Rajashekar ST. Liver function in dengue and its correlation with disease severity: a retrospective cross-sectional observational study in a tertiary care center in Coastal India. Pan Afr Med J. 2021 Dec 23;40:261. doi: 10.11604/pamj.2021.40.261.29795. eCollection 2021. PMID 35251455
- [Result] Thanachartwet V, Desakorn V, Sahassananda D, Jittmittraphap A, Oer-Areemitr N, Osothsomboon S, Surabotsophon M, Wattanathum A. Serum Procalcitonin and Peripheral Venous Lactate for Predicting Dengue Shock and/or Organ Failure: A Prospective Observational Study. PLoS Negl Trop Dis. 2016 Aug 26;10(8):e0004961. doi: 10.1371/journal.pntd.0004961. eCollection 2016 Aug. PMID 27564863
- [Result] Trieu HT, Khanh LP, Ming DKY, Quang CH, Phan TQ, Van VCN, Deniz E, Mulligan J, Wills BA, Moulton S, Yacoub S. The compensatory reserve index predicts recurrent shock in patients with severe dengue. BMC Med. 2022 Apr 7;20(1):109. doi: 10.1186/s12916-022-02311-6. PMID 35387649
- [Result] Yacoub S, Trung TH, Lam PK, Thien VHN, Hai DHT, Phan TQ, Nguyet OPK, Quyen NTH, Simmons CP, Broyd C, Screaton GR, Wills B. Cardio-haemodynamic assessment and venous lactate in severe dengue: Relationship with recurrent shock and respiratory distress. PLoS Negl Trop Dis. 2017 Jul 10;11(7):e0005740. doi: 10.1371/journal.pntd.0005740. eCollection 2017 Jul. PMID 28692675